CLINICAL TRIAL: NCT04606277
Title: The Effect of Smartphone Addiction on Physical Activity and Depression in University Students
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Barış CELBEK, Lecturer, Istanbul Aydın University
Other Study IDs: Barış Celbek, İAU
Record Dates: First submitted 2020-10-24; First posted 2020-10-28 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Young Adult

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young Adult
  Interventions: Other: Smartphone addiction scale, physical activity scale and depression questionnaire

INTERVENTIONS:
Other: Smartphone addiction scale, physical activity scale and depression questionnaire — Telephone addiction of the subjects was measured. Then, physical activity levels were questioned, and finally depression scale was applied.

SUMMARY:
This study was planned considering that young people with smartphone addiction are depressed and their physical activity is significantly reduced. In this direction, our aim is to examine the relationship between smartphone use and physical activity among universities in the 18-25 age group, which uses technology extensively. Our results are to raise awareness of this prevention by uncovering the possibility that it may be the cause of smartphone use in young people.

DETAILED DESCRIPTION:
Smartphone addiction short scale, beck depression questionnaire and international physical activity(IPA) scale short form questionnaires were used in our study.

ELIGIBILITY:
Inclusion Criteria:

1. Being a university student
2. Voluntary participation in the study
3. The adults who were diagnosed as having palliative care needs and are considered to be within the last 5 years of life as determined by their medical practitioner
4. Age between 18-25 years
5. Able to provide consent
6. Have the means to communicate
7. Able to read, understand, and provide informed consent in Turkish

Exclusion Criteria:

1. No chronic wrist deformity or disease
2. Unable to meer the iclusion criteria
3. Too unwell to participate
4. Physical impairments precluding participation in physical activity;
5. Unwilling or unable to sign the Participant Informed Consent Form; Received a diagnosis of brain cancer or thyroid cancer. Brain cancer survivors will be excluded as a function of the cognitive impairments associated with their diagnosis and treatment and thyroid cancer survivors will be excluded due to the vastly different treatment regimens. That is, both of these cancers may result in different physical, psychological/emotional, and social effects that could impact the outcomes of interest.

Eligible participants who want to participate in the other pre-specified outcome measures to assess cognitive functioning must also meet the following additional inclusion/exclusion criteria.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Being a student at the health services vocational school at Istanbul Aydın University
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory | The measurement is one-time and will take 5-10 minutes. It will take an average of 3 weeks after the data of all participants are collected. Then, after 5 months, the evaluation will be completed and the study will be published
  The Beck Depression Inventory (BDI) is widely used to screen for depression and to measure behavioral manifestations and severity of depression. The inventory contains 21 self-report items which individuals complete using multiple choice response formats.
  Depression grade Total
  * Minimal depression 0-9
  * Mild depression 10-16
  * Moderate depression 17-29 Severe depression 30-63
Smartphone Addiction Scale-Short | The measurement is one-time and will take 5-10 minutes. It will take an average of 3 weeks after the data of all participants are collected. Then, after 5 months, the evaluation will be completed and the study will be published
  Smartphone addiction scale (SAS) is a scale for smartphone addiction that consisted of 6 factors and 33 items with a six-point Likert scale (1: "strongly disagree" and 6: "strongly agree") based on self-reporting.Scale items It was scored from 1 to 6. Scale scores range between 10-60. Obtained from the test the higher the score, the higher the risk for addiction are evaluated. The scale has one factor and they do not have scales. For men in the Korean sample The cut-off point was determined as 31, and 33 for women.
International Physical Activity Questionnaire | The measurement is one-time and will take 5-10 minutes. It will take an average of 3 weeks after the data of all participants are collected. Then, after 5 months, the evaluation will be completed and the study will be published
  International Physical Activity Questionnaire Short form (7 questions); gait, moderate to severe information about time spent on activities and time spent sitting provides. Calculation of the total score for the short form is based on walking, moderate activity and It includes the total duration (minutes) and frequency (days) of the activity. For activities The energy required is calculated by the MET-minute score. Standard MET for these activities values were established.
  Seating 1.5 MET Walking 3.3 MET Moderate Physical Activity 4.0 MET Severe Physical Activity 8.0 MET

CONTACTS AND LOCATIONS:
Locations (1):
- Barış CELBEK, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No